CLINICAL TRIAL: NCT04500522
Title: Vaginal Isonicotinic Acid Hydrazide (INH) Prior to Diagnostic Office Hysteroscopy in Primarily Infertile Patients: a Randomized Controlled Trial
Brief Title: Vaginal Isonicotinic Acid Hydrazide Prior to Diagnostic Office Hysteroscopy in Primarily Infertile Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/355/4/19
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Isoniazid

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 vaginal tablet of isonicotinic acid hydrazide (INH) 900 mg inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: INH
- Placebo Comparator (Placebo Comparator): 3 vaginal tablet of Placebo inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INH — 3 vaginal tablet of isonicotinic acid hydrazide 900 mg inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Other Names: isonicotinic acid hydrazide
  Arms: INH
Drug: Placebo — 3 vaginal tablet of Placebo inserted by the patient 12 hours before the scheduled office hysteroscopy.
  Arms: Placebo Comparator

SUMMARY:
To compare the effectiveness of vaginal isonicotinic acid hydrazide with placebo in minimizing the pain experienced by primarily infertile patients during diagnostic ofﬁce hysteroscopy and to assess the ease of insertion of hysteroscope as reported by the hysteroscopist.

DETAILED DESCRIPTION:
hysteroscopy is commonly used in the diagnosis and treatment of intrauterine lesions such as polyps, ﬁbroids, septa, and adhesions, and in the presence of abnormal bleeding and during the removal of an intrauterine device or foreign body. Cervical ripening is made possible by the use of medication through different routes.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women with primary infertility requiring a diagnostic hysteroscopy as a part of an infertility diagnosis workup

Exclusion Criteria:

* women with suspected pregnancy
* heavy vaginal bleeding
* recent pelvic infection
* those known to have hypersensitivity or contraindication to isonicotinic acid hydrazide
* those who received analgesics prior to office heavy vaginal bleeding
* recent pelvic infection
* a concomitant neurologic disease that could affect the correct evaluation of pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — nulliparous women with primary infertility
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores | 10 minutes
  Pain intensity will be assessed by visual analogue scale during the procedure. visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Intensity of pain | 30 minutes after the procedure
  Pain intensity will be assessed by visual analogue scale 30 minutes after the procedure.visual analogue scale ranging from 0 to 10
Operative time | 15 minutes
  From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No